CLINICAL TRIAL: NCT05737810
Title: Attitudes and Unmet Needs Among Type 2 Diabetes Patients
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-7687; U1111-1286-0886 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with Type 2 Diabetes: Participants are recruited via email through online panel companies
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The main purpose of this study is to explore experiences and understand the unmet needs of people with Type 2 Diabetes (T2D) among those who are being managed with basal insulin and those who are insulin naïve in order to understand perspectives for a once weekly insulin option; including any potential barriers to being managed with insulin therapy overall. Study participants will be recruited to complete a 15-minute self-administered online survey.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, age above or equal between 18 to 65 years at the time of signing informed consent.
3. Diagnosed with T2D and currently treating T2D with at least one medication
4. Insulin user that is not using insulin pump
5. Lives in a target country

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
3. Does not meet inclusion criteria requirements

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The main purpose of this study is to explore experiences and understand the unmet needs of people with Type 2 Diabetes among those who are being managed with basal insulin and those who are insulin naïve in order to understand perspectives for a once weekly insulin option; including any potential barriers to being managed with insulin therapy overall.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Current medication burden | At the time of survey response (Day1)
  Numerical; Multiple select from defined list
Injection perceptions | At the time of survey response (Day1)
  Likert scale for measurement of agreement from 1 "strongly disagree" to 7 "strongly agree"
Attitudes regarding T2D overall | At the time of survey response (Day1)
  Likert scale for measurement of agreement from 1 "strongly disagree" to 7 "strongly agree"
Attitudes regarding T2D treatment | At the time of survey response (Day1)
  Likert scales for measurement of satisfaction from 1 "extremely unsatisfied" to 7 "extremely satisfied" and agreement from 1 "strongly disagree" to 7 "strongly agree"
Attitudes regarding insulin icodec | At the time of survey response (Day1)
  Likert scales for measurement of likelihood from 0 "not at all likely" to 10" extremely likely" and agreement from 1 "strongly disagree" to 7 "strongly agree; Rank top 3 from defined list

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (7):
- Novo Nordisk Investigational Site, Sydney, Australia
- Novo Nordisk Investigational Site, Chartres, France
- Novo Nordisk Investigational Site, Bengaluru, India
- Novo Nordisk Investigational Site, Mexico City, Mexico
- Novo Nordisk Investigational Site, Riyadh, Saudi Arabia
- Novo Nordisk Investigational Site, Seoul, South Korea
- Novo Nordisk Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com